CLINICAL TRIAL: NCT02462863
Title: Treatment of Type 2 Diabetes With Immunonutrients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Christ Hospital (Other)
Collaborators: Shriners Hospitals for Children (Other); University of Cincinnati (Other)
Responsible Party: Principal Investigator, Linda H. Martin, RN, BSN, MBA,, MD, The Christ Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-6677
Record Dates: First submitted 2015-05-28; First posted 2015-06-04 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; fish oil; arginine; hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperglycemia | interventions — Arginine; Fish Oils

STUDY DESIGN:
Intervention Model Description: subjects will take arginine 4.5 grams BID plus Fish Oil 7 grams daily
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immunonutrient treatment (Experimental): Administration of arginine and fish oil.
  Interventions: Dietary Supplement: Arginine and fish oil

INTERVENTIONS:
Dietary Supplement: Arginine and fish oil — Dietary supplements

SUMMARY:
The purpose of this research study is to determine if the nutrients arginine and fish oil will reverse or improve diabetes and to find out what additional good or bad effects a combination of arginine and fish oil may have. Both arginine and fish oil are common nutrients taken by normal people on a frequent basis. However, they have not been used in combination in the proposed doses to reverse diabetes once it is established. This study has been approved by the Food and Drug Administration (FDA investigational new drug [IND] 12191).

DETAILED DESCRIPTION:
The hypothesis for the proposed studies is that selected immunonutrients will reduce glucose levels in type 2 diabetes and provide the basis for safe and effective treatment. This should result in an increased resistance to infection, decrease in cardiovascular disease and improve mortality as will be shown in subsequent studies.

Specific Aim 1: To demonstrate proof of concept that supplementation of a normal (diabetic) diet with oral arginine and fish oil will reverse or at least improve glucose control, and improve hemoglobin A1c (HgA1c) in patients with type 2 diabetes.

Specific Aim 2: To determine the relationship of plasma amino acid profiles and concentration of selected fatty acids in cellular (RBC) membranes to the resolution of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adult onset diabetics, BMI under 35 with stable glycemic and hypertensive control. Must be receiving medication for diabetes, be free of cardiac problems such as myocardial infarction, atrial fibrillation or flutter, severe hepatic or gastrointestinal disease, and have a glomerular filtration rate (GFR) of greater than 50 ml/minute. Must have an LDL-C of less than 120 mg/ml with or without treatment.

Exclusion Criteria:

* Chronic infection, past history of cancer except cured skin cancer. Active inflammation processes will also be excluded. Pregnant or nursing women will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
Improvement of type 2 diabetes | 6 months
  Decrease in hemoglobin A1c and glucose.

CONTACTS AND LOCATIONS:
Overall Officials: J. Wesley Alexander, M.D., Sc.D., Principal Investigator — University of Cincinnati; Meenakshi Iyer, M.D., Principal Investigator — The Christ Hospital
Locations (1):
- J. Wesley Alexander, M.D., Sc.D., Cincinnati, Ohio, United States